CLINICAL TRIAL: NCT02567032
Title: Mechanisms and Effects of Oxytocin on Social Cognition in Schizophrenia - Behavioral
Brief Title: Adult Study Oxytocin - Behavioral
Acronym: ASO-Behavioral
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Joshua Woolley, Principal Investigator, University of California, San Francisco
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 10-02262
Record Dates: First submitted 2015-09-29; First posted 2015-10-02 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Schizophrenia; Oxytocin; Social Cognition; Psychotic Disorders
Keywords: Oxytocin; Syntocinon; Social Cognition; Schizophrenia; Psychosis; Schizoaffective Disorder; Schizophreniform Disorder; Psychotic Disorders
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Experimental): 40 IU Oxytocin
  Interventions: Drug: Oxytocin
- Saline Nasal Spray (Placebo Comparator): Placebo Comparator
  Interventions: Drug: Saline Nasal Spray

INTERVENTIONS:
Drug: Oxytocin — 40 IU of the oxytocin will be administered intranasally for a one time dose at the beginning of the visit.
  Other Names: Syntocinon
  Arms: Oxytocin
Drug: Saline Nasal Spray — 40 IU of the saline nasal spray will be administered once at the beginning of the visit.
  Other Names: Placebo
  Arms: Saline Nasal Spray

SUMMARY:
In this study, investigators will examine the behavioral effects and neurophysiological mechanisms of the pro-social neuropeptide oxytocin in patients with recent-onset schizophrenia and other psychotic disorders. Such research is a necessary first step towards identifying whether intranasal oxytocin administration can serve as an adjunct treatment for social impairments in schizophrenia and other psychotic disorders.

Aim 1: To quantify the effects of exogenous oxytocin on social cognition and behavior in patients with recent-onset schizophrenia.

Hypothesis A: Patients and healthy comparison subjects will show enhanced social cognition (e.g., improved interpretation of paralinguistic and emotional cues, such as those involved in emotional or sarcastic communication) after administration of oxytocin versus placebo.

Hypothesis B: Patients and healthy comparison subjects will show increased attention to others' eyes and patients will exhibit increased facial affect expressivity after administration of oxytocin versus placebo.

DETAILED DESCRIPTION:
Part 2: A supplementary study will be added to the proposed parent study, which includes additional behavioral testing consisting of several social cognition computer tasks, clinical assessments, physiological measurements, and questionnaires. The study will be conducted with the same study arms and study interventions as in the proposed parent study. For this supplementary study, the inclusion criteria has broadened to include patients with bipolar disorder with psychotic features and brief psychotic disorder.

ELIGIBILITY:
Inclusion Criteria for Patients:

* 18 to 45 years of age
* Clinically stable
* English Speaking
* Meet DSM-5 criteria for schizophrenia, schizophreniform, schizoaffective disorder, bipolar disorder with psychotic features, or brief psychotic disorder
* No or at most only minor changes to medications in the past week
* Able to use nasal spray
* Must be capable of providing informed consent

Inclusion Criteria for healthy volunteers:

* 18 to 45 years of age
* Clinically stable
* English Speaking
* No diagnosis of mental disorder according to DSM-5, not including mild alcohol use disorder or mild cannabis use disorder
* Able to use nasal spray
* Must be capable of providing informed consent

Exclusion Criteria for Patients:

* Active substance and alcohol use disorder in the past month as determined by the DSM-5 criteria, not including cannabis use disorder
* Subjects with atrophic rhinitis, recurrent nose bleeds, severe brain trauma, and cranial-surgical procedures (hypophysectomy)
* Medical conditions like congestion or sinus problems that could interfere with the study as per the opinion of the investigator
* Hearing deficits
* Pregnancy
* Severe brain trauma

Exclusion Criteria for Healthy Controls:

* Active substance and moderate/severe alcohol use disorder, or mood disorder in the past month as determined by the DSM-5 criteria, not including mild alcohol use disorder or mild cannabis use disorder
* Meet for a current psychiatric disorder according to DSM-5 criteria
* Subjects with atrophic rhinitis, recurrent nose bleeds, severe brain trauma, and cranial-surgical procedures (hypophysectomy)
* Medical conditions like congestion or sinus problems that could interfere with the study as per the opinion of the investigator
* Hearing deficits
* Pregnancy
* Severe brain trauma

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 324 (Actual)
Dates: Start 2010-10; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Change in Social Cognition Task Performance | Through study completion, 2-3 weeks
  Participants will undergo computer tasks that measure social cognition. Tasks will involve verbal responses, pressing buttons at specific times, listening, and viewing audio-visual stimuli. Investigators will be measuring the difference in accuracy and verbal content of the responses on the oxytocin day compared to the placebo day.

SECONDARY OUTCOMES:
Physiological Measurements | Through study completion, 2-3 weeks
  Sensors will be attached to measure heart rate, respiration, and skin conductance during computer tasks.
Questionnaire | At baseline visit, up to 4 hours
  Participants will be asked questions about their current positive and negative symptoms, medical and psychiatric history. Self-report responses will be saved in writing or audio recording.

CONTACTS AND LOCATIONS:
Overall Officials: Josh D Woolley, MD/PhD, Principal Investigator — University of California San Francisco, San Francisco Veterans Affairs Medical Center
Locations (2):
- United States (2):
  - San Francisco Veterans Affairs Medical Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California